CLINICAL TRIAL: NCT04391452
Title: Effect of a Dietary Supplement Based on Magnesium, Vitamins, Rhodiola and L-theanine (Stress Resist®), on Stress in Stressed Subjects: Randomized Study Versus Placebo.
Brief Title: Dietary Supplement With Magnesium, Vitamins, Rhodiola and L-theanine Stressed Subjects: Randomized Study Versus Placebo (MAGRITTE)
Acronym: MAGRITTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBHP 2019 PICKERING 3; 2020-A00040-39 (Other: ANSM)
Record Dates: First submitted 2020-04-21; First posted 2020-05-18 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2020-04

CONDITIONS: Stress, Psychological
Keywords: Stressed individuals; Dietary supplement; Magnesium; fMRI
MeSH Terms: conditions — Stress, Psychological | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: After pre-selection (Day-14 to Day 0), participants will receive one of the two products in random order (Mg or placebo).
  Treatment allocation will follow a randomization plan and will be carried out by a Clinical Research Associate totally independent from the protocol. The randomization list and a copy will be edited, placed in a sealed envelope, and submitted to the Pharmacy of the University Hospital of Clermont-Ferrand and the Clinical Pharmacology Centre of Clermont-Ferrand which is the coordinating centre.
  For a 5% risk of bilateral species error and a 90% power, it is necessary to include 50 subjects per group to highlight such an effect size. In addition, fMRI examinations will be offered to the first 20 subjects included per group, i.e. 40 subjects, an usual and relatively consensual number for fMRI work.
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement group (Experimental): Group 1:50 stressed subjects who will have a 28-day intake of dietary supplement. Of the 50 stressed subjects, 20 subjects will participate in the fMRI exam. Dietary supplement is composed of Mg (150 mg), Vitamin B6 (0.7 mg), Vitamin B9 (100µg), Vitamin B12 (1.25 µg), rhodiola (222mg), and green tea/L-théanine (125 mg).
  Interventions: Dietary Supplement: Stress Resist® (oral dietary supplement)
- Placebo group (Placebo Comparator): Group 2 (Placebo comparator (lactose)): 50 stressed subjects who will have a 28-day intake of placebo. Of the 50 stressed subjects, 20 subjects will participate in the fMRI exam.
  Interventions: Dietary Supplement: Stress Resist® (oral dietary supplement)

INTERVENTIONS:
Dietary Supplement: Stress Resist® (oral dietary supplement) — Stress Resist® (dietary supplement) is composed of Mg (150 mg), Vitamin B6 (0.7 mg), Vitamin B9 (100µg), Vitamin B12 (1.25 µg), rhodiola (222mg), and green tea/L-théanine (125 mg). Oral supplementation. All subjects in the MAGRITTE study will receive either a dietary supplement or a placebo for 28 days (morning intake). The effects on stress will be studied both with questionnaires, biological samples (blood, urine and stool), with a Heart Rate Variability test. 40 subjects (20 subjects per group) will have an fMRI exam.

SUMMARY:
The aim is to study the effect of a dietary supplement on stress and pain through questionnaires and follow-up of physiological parameters, and functional Magnetic Resonance Imaging (fMRI) in stressed healthy subjects versus stressed healthy subjects without treatment.

DETAILED DESCRIPTION:
The MAGRITTE monocentric study conducted at Clermont-Ferrand University Hospital is a parallel, randomized, and controlled versus placebo performed in stressed subjects.

The main outcome of this study is to demonstrate on stress the effectiveness of a dietary supplement based on magnesium (Mg), vitamins, rhodiola and L-Theanine, compared to placebo, in subjects with chronic stress and free from other pathologies.

The secondary objectives are to evaluate the action of Mg dietary supplement on:

1. pain by the Numerical Scale and fMRI,
2. stress by the Numerical Scale and fMRI,
3. anxiety, depression and sleep with questionnaires,
4. selected biological parameters,
5. heart rate variability,
6. microbiota,
7. safety of the product.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 65,
* Subject with stress (DASS-42 screening scale ≥14) and having been under stress for at least 1 month,
* Subject free of any introduction of new treatment or diet at the time inclusion,
* Subject free of any treatment in the 7 days prior to inclusion including no use of analgesic or anti-inflammatory drugs,
* Cooperation and understanding sufficient to comply with the requirements of the study,
* Acceptance to give written consent,
* Affiliation with the French Social Security,
* Registration or acceptance of registration in the national register of volunteers participating in Research.

Exclusion Criteria:

* Contraindications to the realization of MRI without injection such as claustrophobia proven, hearing aid, pacemaker wearers, wearing a brain clip,
* Contraindication to Mg administration: hypersensitivity to Mg oxide, or to one of the excipients,
* With magnesemia > 1.07 mmol/l,
* With moderate (or more severe) kidney failure with creatinine clearance <60 ml/min,
* Receiving a treatment or dietary supplement containing Mg, pre- or probiotics, or herbal extracts (e.g. anti-stress, anti-inflammatory, analgesic) at the time of inclusion,
* Treated with antibiotics in the three months prior to inclusion,
* Having a medical and/or surgical history judged by the investigator or his or her representative that are not compatible with the trial,
* Evolutionary pathology at the time of the inclusion,
* Excessive consumption of alcohol, tobacco (up to 10 cigarettes per day), coffee, tea or drink containing caffeine (equivalent to more than 4 cups per day) or substance abuse,
* Subject who does not meet the selection criteria for their ability to discriminate against sensations resulting from nociceptive stimulation during psychometric tests,
* Subject who does not meet the selection criteria for their ability to discriminate against colours projected during the fMRI exam,
* Subject participating in another clinical trial, or in the exclusion period, or having received a total amount of compensation of more than 4,500 euros over the 12 months prior to the start of the trial,
* Woman of childbearing age not using an effective contraceptive method, pregnant woman or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Measure of stress with DASS-42 | Day 0
  The measure of stress with stress subscale in magnesium and placebo groups will be performed in order to assess the impact of the dietary supplement on this parameter. This subscale consists of 14 questions of self-evaluation, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of stress
Measure of the impact of a dietary supplement (based on Mg, vitamins, rhodiola and L-Theanine) on stress with DASS-42 after 28 days of treatment | Day 28
  The measure of stress with stress subscale in magnesium and placebo groups will be performed in order to assess the impact of the dietary supplement on this parameter. This subscale consists of 14 questions of self-evaluation, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of stress

SECONDARY OUTCOMES:
Impact of a dietary supplement on pain induced by thermal stimulation observed by fMRI | Day 28
  Pain intensity will be assessed by the numerical pain rating scale (NPRS): the scale ranges from 0 "no pain" to 10 "maximal tolerable pain" following different thermal stimulations (using Pathway Medoc®) applied in fMRI
Impact of a dietary supplement on pain induced by thermal stimulation observed by fMRI | Day 0
  Pain intensity will be assessed by the numerical pain rating scale (NPRS): the scale ranges from 0 "no pain" to 10 "maximal tolerable pain" following different thermal stimulations (using Pathway Medoc®) applied in fMRI
Impact of dietary supplement on pain matrix observed by fMRI | Day 0
  Integration will be measured by BOLD signal at the pain matrix (primary and secondary somatosensory cortex, insular cortex, cingulate cortex prefrontal cortex and Basal Ganglia).
Impact of dietary supplement on pain matrix observed by fMRI | Day 28
  Integration will be measured by BOLD signal at the pain matrix (primary and secondary somatosensory cortex, insular cortex, cingulate cortex prefrontal cortex and Basal Ganglia).
Evaluation of the analgesic effect of dietary supplement during the period of 28 days of treatment | Over the period of treatment : Day 0 to Day 28
  A daily pain diary will be given to patients for the 28 days of treatment in order to score their average pain during this period. Pain intensity will be assessed by the NPRS obtained from the daily pain diary: the scale ranges from 0 "no pain" to 10 "maximal tolerable pain".
Impact of dietary supplement on stress by DASS-42 questionnaire | Day 0
  Stress will be measured by DASS-42 questionnaire in dietary supplement and placebo groups. This subscale consists of 14 questions of self-evaluation Depression Anxiety Stress Scale-42, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of stress
Impact of dietary supplement on stress by DASS-42 questionnaire | Day 14
  Stress will be measured by DASS-42 questionnaire in dietary supplement and placebo groups. This subscale consists of 14 questions of self-evaluation Depression Anxiety Stress Scale-42, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of stress
Impact of dietary supplement on stress by DASS-42 questionnaire | Day 28
  Stress will be measured by DASS-42 questionnaire in dietary supplement and placebo groups. This subscale consists of 14 questions of self-evaluation Depression Anxiety Stress Scale-42, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of stress
Impact of dietary supplement on stress by DASS-42 questionnaire | Day 56
  Stress will be measured by DASS-42 questionnaire in dietary supplement and placebo groups. This subscale consists of 14 questions of self-evaluation Depression Anxiety Stress Scale-42, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of stress
Effect of dietary supplement on increased stress induced by visual stimulation | Day 0
  Stress intensity will be assessed by the numerical stress rating scale: the scale ranges from 0 "no stress" to 10 "maximal stress" following different visual stimulation induced by different colors during the anticipatory phase in fMRI.
Effect of dietary supplement on increased stress induced by visual stimulation | Day 28
  Stress intensity will be assessed by the numerical stress rating scale: the scale ranges from 0 "no stress" to 10 "maximal stress" following different visual stimulation induced by different colors during the anticipatory phase in fMRI.
Evaluation of the stress effect of dietary supplement by numerical scale during the period of 28 days of treatment | Over the period of treatment: Day 0 to Day 28
  Stress intensity will be assessed by the numerical stress rating scale: the scale ranges from 0 "no stress" to 10 "maximal stress" during the ratings framing the fMRI exam before and after taking a dietary supplement.
Evaluation of the stress effect of dietary supplement by numerical scale | Day 28
  Stress intensity will be assessed by the numerical stress rating scale: the scale ranges from 0 "no stress" to 10 "maximal stress" during the ratings framing the fMRI exam before and after taking a dietary supplement.
Impact of dietary supplement on stress matrix observed by fMRI | Day 0
  Integration difference will be measured by bold signal at the stress matrix level (hippocampus, prefrontal cortex, amygdala and basal ganglia)
Impact of dietary supplement on stress matrix observed by fMRI | Day 28
  Integration difference will be measured by bold signal at the stress matrix level (hippocampus, prefrontal cortex, amygdala and basal ganglia)
Evaluation of stress level by daily diary | Day 0
  Stress level will be observed over 28 days of treatment from the daily diary data using a numerical stress scale: scores ranging from 0 "no stress" to 10 "maximal stress".
Evaluation of stress level by daily diary | Day 28
  Stress level will be observed over 28 days of treatment from the daily diary data using a numerical stress scale: scores ranging from 0 "no stress" to 10 "maximal stress".
Effect of dietary supplement on anxiety | day 0
  Anxiety will be measured by DASS-42 questionnaire in dietary supplement and placebo groups. This subscale consists of 14 questions of self-evaluation Depression Anxiety Stress Scale-42, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of anxiety.
Effect of dietary supplement on anxiety | day 14
  Anxiety will be measured by DASS-42 questionnaire in dietary supplement and placebo groups. This subscale consists of 14 questions of self-evaluation Depression Anxiety Stress Scale-42, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of anxiety.
Effect of dietary supplement on anxiety | day 28
  Anxiety will be measured by DASS-42 questionnaire in dietary supplement and placebo groups. This subscale consists of 14 questions of self-evaluation Depression Anxiety Stress Scale-42, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of anxiety.
Effect of dietary supplement on anxiety | day 56
  Anxiety will be measured by DASS-42 questionnaire in dietary supplement and placebo groups. This subscale consists of 14 questions of self-evaluation Depression Anxiety Stress Scale-42, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of anxiety.
Evaluation of the effect of dietary supplement on depression | day 0
  Depression will be measured by DASS-42 questionnaire in dietary supplement and placebo groups. This subscale consists of 14 questions of self-evaluation Depression Anxiety Stress Scale-42, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of depression
Evaluation of the effect of dietary supplement on depression | day 14
  Depression will be measured by DASS-42 questionnaire in dietary supplement and placebo groups. This subscale consists of 14 questions of self-evaluation Depression Anxiety Stress Scale-42, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of depression
Evaluation of the effect of dietary supplement on depression | day 28
  Depression will be measured by DASS-42 questionnaire in dietary supplement and placebo groups. This subscale consists of 14 questions of self-evaluation Depression Anxiety Stress Scale-42, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of depression
Evaluation of the effect of dietary supplement on depression | day 56
  Depression will be measured by DASS-42 questionnaire in dietary supplement and placebo groups. This subscale consists of 14 questions of self-evaluation Depression Anxiety Stress Scale-42, each of them emphasizing a negative emotional symptom, these feelings of uselessness and hopelessness. Each element is evaluated from zero to three, zero being "not present" and three being "very frequently". It assesses mental health by measuring the severity of depression
Evaluation of the effect of the dietary supplement on quality of sleep | day 0
  The Pittsburg Sleep Questionnaire Index is a self-questionnaire including 19 items. It was developed to measure the quality of sleep over the month before the patient interview. This questionnaire includes 7 components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, hypnotic medication use and daytime dysfunction. In scoring the PSQI, seven component are evaluated from 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality. A score > 5 indicates a sleep disturbance.
Evaluation of the effect of the dietary supplement on quality of sleep | day 14
  The Pittsburg Sleep Questionnaire Index is a self-questionnaire including 19 items. It was developed to measure the quality of sleep over the month before the patient interview. This questionnaire includes 7 components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, hypnotic medication use and daytime dysfunction. In scoring the PSQI, seven component are evaluated from 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality. A score > 5 indicates a sleep disturbance.
Evaluation of the effect of the dietary supplement on quality of sleep | day 28
  The Pittsburg Sleep Questionnaire Index is a self-questionnaire including 19 items. It was developed to measure the quality of sleep over the month before the patient interview. This questionnaire includes 7 components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, hypnotic medication use and daytime dysfunction. In scoring the PSQI, seven component are evaluated from 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality. A score > 5 indicates a sleep disturbance.
Evaluation of the effect of the dietary supplement on quality of sleep | day 56
  The Pittsburg Sleep Questionnaire Index is a self-questionnaire including 19 items. It was developed to measure the quality of sleep over the month before the patient interview. This questionnaire includes 7 components: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, hypnotic medication use and daytime dysfunction. In scoring the PSQI, seven component are evaluated from 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality. A score > 5 indicates a sleep disturbance.
Evaluation of the dietary supplement on catastrophism | day 0
  Pain Catastrophizing Scale (PCS) is a questionnaire in which the patient is asked to describe the kind of thought and emotions they feel during pain. This questionnaire consists of 13 items describing different thoughts or emotions that may be associated with the pain. The patient will have to indicate how much he has these thoughts or emotions when he feels pain by giving a score between 0 and 4, 0: not at all, 4: all the time. The final score is the sum of the scores for each question.
Evaluation of the dietary supplement on catastrophism | day 14
  Pain Catastrophizing Scale (PCS) is a questionnaire in which the patient is asked to describe the kind of thought and emotions they feel during pain. This questionnaire consists of 13 items describing different thoughts or emotions that may be associated with the pain. The patient will have to indicate how much he has these thoughts or emotions when he feels pain by giving a score between 0 and 4, 0: not at all, 4: all the time. The final score is the sum of the scores for each question.
Evaluation of the dietary supplement on catastrophism | day 28
  Pain Catastrophizing Scale (PCS) is a questionnaire in which the patient is asked to describe the kind of thought and emotions they feel during pain. This questionnaire consists of 13 items describing different thoughts or emotions that may be associated with the pain. The patient will have to indicate how much he has these thoughts or emotions when he feels pain by giving a score between 0 and 4, 0: not at all, 4: all the time. The final score is the sum of the scores for each question.
Evaluation of the dietary supplement on catastrophism | day 56
  Pain Catastrophizing Scale (PCS) is a questionnaire in which the patient is asked to describe the kind of thought and emotions they feel during pain. This questionnaire consists of 13 items describing different thoughts or emotions that may be associated with the pain. The patient will have to indicate how much he has these thoughts or emotions when he feels pain by giving a score between 0 and 4, 0: not at all, 4: all the time. The final score is the sum of the scores for each question.
Evaluation of blood Magnesium (Mg) level | day 0
  The intracellular magnesium concentrations will be determined by the blood samples taken
Evaluation of blood Magnesium (Mg) level | day 14
  The intracellular magnesium concentrations will be determined by the blood samples taken
Evaluation of blood Magnesium (Mg) level | day 28
  The intracellular magnesium concentrations will be determined by the blood samples taken
Evaluation of blood Magnesium (Mg) level | day 56
  The intracellular magnesium concentrations will be determined by the blood samples taken
Evaluation of erythrocyte Mg level | day 0
  The erythrocyte magnesium concentrations will be determined by the blood samples taken
Evaluation of erythrocyte Mg level | day 14
  The erythrocyte magnesium concentrations will be determined by the blood samples taken
Evaluation of erythrocyte Mg level | day 28
  The erythrocyte magnesium concentrations will be determined by the blood samples taken
Evaluation of erythrocyte Mg level | day 56
  The erythrocyte magnesium concentrations will be determined by the blood samples taken
Evaluation of urinary Mg level | day 0
  The urinary concentration of magnesium will be determined by the urine collected for 24 hours.
Evaluation of urinary Mg level | day 14
  The urinary concentration of magnesium will be determined by the urine collected for 24 hours.
Evaluation of urinary Mg level | day 28
  The urinary concentration of magnesium will be determined by the urine collected for 24 hours.
Evaluation of urinary Mg level | day 56
  The urinary concentration of magnesium will be determined by the urine collected for 24 hours.
Evaluation of salivary cortisol level | day 0
  The concentration of cortisol will be determined by salivary cortisol dosage and will be performed before and after fMRI exam.
Evaluation of salivary cortisol level | day 28
  The concentration of cortisol will be determined by salivary cortisol dosage and will be performed before and after fMRI exam.
Evaluation of Heart Rate Variability | day 0
  Heart rate variability (HRV / HRV) is a measure of changes in heart rate that will provide an estimate of stress. It is usually calculated by analyzing time series of beat-by-beat intervals of the electrocardiogram or blood pressure plots (using Codesna®).
Evaluation of Heart Rate Variability | day 14
  Heart rate variability (HRV / HRV) is a measure of changes in heart rate that will provide an estimate of stress. It is usually calculated by analyzing time series of beat-by-beat intervals of the electrocardiogram or blood pressure plots (using Codesna®).
Evaluation of Heart Rate Variability | day 28
  Heart rate variability (HRV / HRV) is a measure of changes in heart rate that will provide an estimate of stress. It is usually calculated by analyzing time series of beat-by-beat intervals of the electrocardiogram or blood pressure plots (using Codesna®).
Analysis of the microbiota (stool samples) | day 0
  The stool samples will assess to identify the bacterial biodiversity by a genetic sequencing analysis of bacterial DNA.
Analysis of the microbiota (stool samples) | day 28
  The stool samples will assess to identify the bacterial biodiversity by a genetic sequencing analysis of bacterial DNA.
Assessment of the occurrence of adverse event | day 28
  The adverse event will be reported by the patient on his daily diary during the period of treatment, over 28 days.
Assessment of analgesic consumption | Day 28
  Analgesic consumption will be assessed by the daily diary during the period of treatment, over 28 days
Influence on microbiota assessed by a food survey | Day 28
  A food survey will be performed by the daily diary during the period of treatment, over 28 days. Participant will have to report in his daily diary what he will have eaten per day (breakfast, lunch and dinner).

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pickering, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France